CLINICAL TRIAL: NCT03793712
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled, Fixed-flexible-dose Study of Lu AF11167 for the Treatment of Persistent Prominent Negative Symptoms in Patients With Schizophrenia
Brief Title: Study With Lu AF11167 for the Treatment of Negative Symptoms in Patients With Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy based on interim analysis
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17972A
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lu AF11167 low dose (Experimental)
  Interventions: Drug: Lu AF11167 (1-2 mg/day)
- Lu AF11167 high dose (Experimental)
  Interventions: Drug: Lu AF11167 (3-4 mg/day)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AF11167 (1-2 mg/day) — Fixed-flexible oral dose, tablets. Once daily. 12 weeks.
  Arms: Lu AF11167 low dose
Drug: Lu AF11167 (3-4 mg/day) — Fixed-flexible oral dose, tablets. Once daily. 12 weeks.
  Arms: Lu AF11167 high dose
Drug: Placebo — Placebo oral dose, tablets. Once daily. 12 weeks.
  Arms: Placebo

SUMMARY:
A study to evaluate the efficacy of 2 fixed-flexible doses of Lu AF11167 on negative symptoms in patients with schizophrenia

ELIGIBILITY:
Inclusion Criteria

* The patient has schizophrenia, diagnosed according to DSM-5® as confirmed by the Mini-International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorders Studies (MINI-Schz).
* The patient has been known to the site or investigator and treated by the site or investigator for at least the last 6 months prior to Screening Visit 1.
* The patient has suffered from persistent prominent negative symptoms for the last 6 months prior to the Screening Visit 1, in the opinion of the investigator and recorded in medical records.
* The patient has been treated for schizophrenia with stable doses of an oral antipsychotic within the approved dose range and without any dose increase during the last 6 months prior to Screening Visit 1 (dose reductions are acceptable). Combination therapy of two antipsychotics is only allowed with the written approval of the Medical Monitor in cases where the second antipsychotic is a low-potency first generation antipsychotic drug (e.g., chlorpromazine, promazine or chlorprothixene at low doses) or quetiapine at a dose of ≤150 mg, given in the evening for sleep problems and where both can be discontinued during the washout phase without endangering the patient's safety. Both antipsychotics will be withdrawn during the washout phase and need to be discontinued before Screening Visit 2. Combination therapy of more than 2 antipsychotic medications is not allowed during the previous 6 months prior to Screening Visit 1.
* The patient has had no psychiatric admissions/hospitalization due to a clinical deterioration during the last 6 months prior to Screening Visit 1, this excludes ambulatory visits to ask for advice from the psychiatry team.Patients hospitalized during the last 6 months for social reasons only or patients who are currently hospitalized for social reasons can be included with the Medical Monitor's approval.
* The patient is in a clinically stable phase of schizophrenia and has not more than moderate severity on relevant positive symptoms, that is a score of ≤4 (moderate) out of score of 7 on each of the following PANSS items: Delusions (P1), Hallucinatory behaviour (P3), Suspiciousness / persecution (P6), Uncooperativeness (G8), Unusual thought content (G9) at Screening Visit 1, Washout Visit(s), Screening Visit 2, and Baseline Visit and a score ≤5 on Conceptual disorganization (P2).
* The patient currently has no clinically significant acute extrapyramidal side effects (acute EPS) or tardive dyskinesia (TD) based upon the protocol-specified clinical examination.
* The patient has prominent negative symptoms as demonstrated by a PANSS Marder Negative Symptom Factor Score (NSFS) ≥20 at Screening Visit 1, Washout Visit(s) and Screening Visit 2. NSFS is the sum of scores of the following PANSS items: Blunted affect (N1), Emotional withdrawal (N2), Poor rapport (N3), Passive/apathetic social withdrawal (N4), Lack of spontaneity & flow of conversation (N6), Motor retardation (G7) and Active social avoidance (G16).
* The patient has a Clinical Global Impression-Schizophrenia Severity of Illness (CGI-SCH-S) overall severity score ≤4 at Screening Visit 1.
* The patient does not currently have a diagnosis of Major Depressive Disorder or have depressive symptoms rated with a total score ≥5 on the Calgary Depression Scale for Schizophrenia (CDSS).
* The patient has no history of violent behaviour for the last 12 months prior to Screening Visit 1.
* The patient has a caregiver or an identified responsible person (for example, partner, family member, social worker, case worker, or nurse) considered reliable by the investigator in providing support to the patient to ensure compliance with study treatment, outpatient visits, and protocol procedures.

Exclusion criteria

* The patient has had an acute exacerbation requiring hospitalization within the last 6 months prior to Screening Visit 1.
* The patient has had an acute exacerbation requiring change in antipsychotic medication (with reference to drug or dose) within the last 6 months prior to Screening Visit 1.
* The patient has a current diagnosis or a history of substance use disorder according to DSM-5® criteria within 6 months prior to Screening Visit 1 with the exception of tobacco, or mild cannabis or mild alcohol use disorder (occasional - but not weekly recreational cannabis use is acceptable). Patients with a positive drug screen test for opiates, methadone, cocaine, amphetamines [including ecstasy], barbiturates, verified by repeated testing, are excluded from the study.
* The patient is at significant risk of harming himself/herself or others in the investigator's opinion.
* The patient has tested positive for hepatitis A virus antibody (anti-HAV IgM), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV). If the anti-HCV test result is positive, but acute/chronic infection is excluded with a negative HCV RNA test patient can be included in the study.
* The patient has tested positive for human immunodeficiency virus (HIV).
* The patient has a present condition that might compromise liver function (for example, alcohol abuse, hepatitis, hepatic insufficiency, cholestasis, haemachromatosis, deficit in alpha 1 antitrypsine, Wilson's Disease, autoimmune diseases, cirrhosis).
* The patient has any other disorder for which the treatment takes priority over treatment of schizophrenia or is likely to interfere with the study treatment or impair treatment compliance.

Other in- and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Change in Negative Symptom Scale (BNSS) total score | from baseline to Week 12
  The BNSS is a brief clinician rating scale, intended to measure negative symptoms. It consists of 13 items organized into 6 subscales: anhedonia, distress, asociality, avolition, blunted affect and alogia. The items score the impairment. Items 1 to 4 are rated from 0 (Normal) to 6 (Extremely severe) and items 5 to 13 are rated from 0 (No impairment) to 6 (Severe deficit). The BNSS total score is calculated by summing the 13 individual items; subscale scores are calculated by summing the individual items within each subscale. Users of the BNSS should have training in psychiatric interview techniques and have clinical experience working with patients with schizophrenia and related psychotic disorders. The BNSS total scores ranges from 0 to 78.

SECONDARY OUTCOMES:
Change in Personal and Social Performance (PSP) score | from baseline to Week 12
  The PSP is a clinician-rated scale designed and validated to measure a patient's current level of social functioning. The PSP consists of 4 items: socially useful activities (including work and study), personal and social relationships, self-care, and disturbing and aggressive behaviours. The 4 items are assessed on a 6-point scale, from absent to very severe. Based on these assessments and their combination, individual scores are converted into a global score ranging from 1 to 100.
Change in Positive and Negative Syndrome Scale (PANSS) total score | from baseline to Week 12
  The PANSS is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS includes 3 sub-scales and 30 items
Change in PANSS Marder Negative Symptom Factor score: negative symptoms | from baseline to Week 12
  The PANSS is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS includes 3 sub-scales and 30 items
Change in PANSS Negative subscale score | from baseline to Week 12
  The PANSS is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS includes 3 sub-scales and 30 items
Change in Clinical Global Impression - Schizophrenia (CGI-SCH-S) negative symptoms score | from baseline to Week 12
  The CGI-SCH is a clinician-rated scale to assess global illness severity and degree of change in patients with schizophrenia. For both the global illness severity and degree of change, the CGI-SCH consists of four different groups of symptoms (positive, negative, cognitive and depressive) and the overall severity of the disorder. The CGI-SCH-S severity of illness category symptoms and overall severity are rated on a 7-point scale ranging from 1 (normal - not ill) to 7 (Among the most severely ill). For the first four ratings (positive, negative, depressive, and cognitive symptoms), the assessment should focus on the severity of symptoms only. Additionally, for 'overall severity' rating, both severity of symptoms and interference with functioning should be considered.
Clinical Global Impression - Schizophrenia (CGI-SCH-DC) negative symptoms score | at Week 12
  The CGI-SCH is a clinician-rated scale to assess global illness severity and degree of change in patients with schizophrenia. For both the global illness severity and degree of change, the CGI-SCH consists of four different groups of symptoms (positive, negative, cognitive and depressive) and the overall severity of the disorder. In the CGI-SCH-DC degree of change category symptoms and overall severity are rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Each single rating (conditions of severity and degree of improvement) and overall ratings of severity and improvement are scored independently and no total score is derived.
CGI-SCH-DC negative symptoms response | at Week 12
  The CGI-SCH is a clinician-rated scale to assess global illness severity and degree of change in patients with schizophrenia. For both the global illness severity and degree of change, the CGI-SCH consists of four different groups of symptoms (positive, negative, cognitive and depressive) and the overall severity of the disorder. In the CGI-SCH-DC degree of change category symptoms and overall severity are rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Each single rating (conditions of severity and degree of improvement) and overall ratings of severity and improvement are scored independently and no total score is derived. Response defined as CGI-SCH-DC negative symptoms = 1 or 2
BNSS response | at Week 12
  The BNSS is a brief clinician rating scale, intended to measure negative symptoms. It consists of 13 items organized into 6 subscales: anhedonia, distress, asociality, avolition, blunted affect and alogia. The items score the impairment. Items 1 to 4 are rated from 0 (Normal) to 6 (Extremely severe) and items 5 to 13 are rated from 0 (No impairment) to 6 (Severe deficit). The BNSS total score is calculated by summing the 13 individual items; subscale scores are calculated by summing the individual items within each subscale. Users of the BNSS should have training in psychiatric interview techniques and have clinical experience working with patients with schizophrenia and related psychotic disorders. The BNSS total scores ranges from 0 to 78. Response criteria defined as 20,30 or 40% decrease in BNSS total score.
Change in PANSS -Positive subscale score | from baseline to Week 12
  The PANSS is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS includes 3 sub-scales and 30 items
Change in Clinical Global Impression - Schizophrenia (CGI-SCH-S) severity of illness overall severity score | from baseline to Week 12
  The CGI-SCH is a clinician-rated scale to assess global illness severity and degree of change in patients with schizophrenia. For both the global illness severity and degree of change, the CGI-SCH consists of four different groups of symptoms (positive, negative, cognitive and depressive) and the overall severity of the disorder. The CGI-SCH-S severity of illness category symptoms and overall severity are rated on a 7-point scale ranging from 1 (normal - not ill) to 7 (Among the most severely ill). For the first four ratings (positive, negative, depressive, and cognitive symptoms), the assessment should focus on the severity of symptoms only. Additionally, for 'overall severity' rating, both severity of symptoms and interference with functioning should be considered.
Clinical Global Impression - Schizophrenia (CGI-SCH-DC) degree of change in overall severity score | at Week 12
  The CGI-SCH is a clinician-rated scale to assess global illness severity and degree of change in patients with schizophrenia. For both the global illness severity and degree of change, the CGI-SCH consists of four different groups of symptoms (positive, negative, cognitive and depressive) and the overall severity of the disorder. In the CGI-SCH-DC degree of change category symptoms and overall severity are rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Each single rating (conditions of severity and degree of improvement) and overall ratings of severity and improvement are scored independently and no total score is derived.
Change in Calgary Depression Scale for Schizophrenia (CDSS) total score | from baseline to Week 12
  The CDSS is a 9-item clinician rated scale specifically developed for the assessment of depression in patients with schizophrenia. The items on the CDSS are all typical depressive symptoms and do not appear to overlap with the negative symptoms of schizophrenia. All items are rated on a 4-point scale from 0 (absent) to 3 (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (53):
- Bulgaria (13):
  - Mental Health Center Prof. Dr. Ivan Temkov EOOD (BG0001), Burgas
  - MHAT Dr. Hristo Stambolski (BG0007), Kazanlak
  - State Psychiatric Hospital Lovech (BG0012), Lovech
  - First Department for men with acute mental diseases-NPH Sv. Ivan Rilski (BG0010), Novi Iskar
  - UMHAT Dr.Georgi Stranski EAD (BG0006), Pleven
  - Dr.Svetlozar Georgiev MD, Office of Office of Ambulatory for Group Practice for Specialized Psychiartic Help ¿ PHILIPOPOLIS OOD (BG0014), Plovdiv
  - State Psychiatric Hospital - Sevlievo (BG009), Sevlievo
  - Medical Center INTERMEDICA (BG0003), Sofia
  - DCC Mladost-M (BG0004), Varna
  - DCC Mladost-M Varna OOD (BG0005), Varna
  - Med Centre Medical plus (BG008), Varna
  - Center for Mental Health Veliko Tarnovo (BG0013), Veliko Tarnovo
  - Mental Health Center-Vratsa EOOD (BG0002), Vratsa
- Czechia (6):
  - Dr.Jan Holan MD, Office of (CZ0003), Brno
  - Meditrine s.r.o. - Psychiatricka Ambulance, Lecebne Centrum (CZ0005), Havířov
  - Clinline services s.r.o. (CZ0006), Hostivice
  - Neuropsychiatrie HK, s.r.o. (CZ0004), Hradec Králové
  - A-Shine s.r.o. (CZ0001), Pilsen
  - Institute of Neuropsychiatric Care (INEP) (CZ0007), Prague
- Estonia (2):
  - Marienthali Kliinik (EE0001), Tallinn
  - OU Jaanson & Laane (EE0002), Tartu
- Germany (5):
  - Medical Pratice For Neurology/Psychiatry (DE0003), Berlin
  - Office of Dr.Kirsten Hahn (DE0002), Berlin
  - Zentralinstitut fur Seelische Gesundheit (ZI)-Leitung Abteilung Molekulares Neuroimaging (DE0004), Mannheim
  - Dr. Frank Kuehn MD, Office Of (DE001), Oranienburg
  - Klinikum der Eberhard-Karls-Universitaet Tuebingen (DE0007), Tübingen
- Hungary (7):
  - Nyiro Gyula Hospital - OPAI (HU0006), Budapest
  - Semmelweis Egyetem-Neurologiai Klinika (HU0005), Budapest
  - Bugat Pal Hospital (HU0008), Gyöngyös
  - Dr Mathe es Tarsa Bt (HU0001), Kalocsa
  - Somogy Megyei Kaposi Mor Oktato Korhaz (HU0003), Kaposvár
  - Szabolcs-Szatmar-Bereg megyei Korhazak es Egyetemi Oktatokorhaz, Josa Andras Oktatokorhaz, Pszichiatriai es Pszichoterapias Osztaly (HU0002), Nyíregyháza
  - Javorszky Odon Hospital (HU0004), Vác
- Latvia (5):
  - Daugavpils Psychoneurological Hospital (LV0005), Daugavpils
  - Hospital Gintermuiza (LV0001), Jelgava
  - Jsc Piejuras Slimnica Psychiatry Clinic (LV0003), Liepāja
  - Riga Centre Of Psychiatry And Addiction Disorders (LV0002), Riga
  - Sigulda Hospital Outpatient Clinic (LV0006), Sigulda
- Poland (6):
  - Gabinet Lekarski Psychiatryczny Ireneusz Kaczorowski (PL0012), Bełchatów
  - Wlokiennicza Med Specjalistyczna Praktyka Lekarska dr n. med. Tomasz Markowski (PL0005), Bialystok
  - Med-Ars (Pl0010), Bydgoszcz
  - Centrum Zdrowia Psychicznego Biomed - Jan Latala (PL0006), Kielce
  - Przychodnia Syntonia Izabela Chojnowska-Cwiakala (PL0011), Kielce
  - Syntonia Sp. z o.o. (PL0002), Pruszcz Gdański
- Ukraine (9):
  - Si Inpn Namsu (Ua0003), Kharkiv
  - Si Inpn Namsu (Ua0008), Kharkiv
  - Kherson Regional Psychiatric Hospital (UA0009), Kherson
  - Kiev Regional Specialized Psycho-Narcological Medical Care (UA0005), Kiev
  - Communal Institution Kirovograd Regional Psychiatric Hospital. Donetsk National Medical University, Chair of psychiatry, psychotherapy, narcology and medical psychology (UA0004), Kropyvnytskyi
  - Railway Clinical Hospital #1, Ukr Research Institute, Social And Forensic Psychatriy And Drug Abuse (UA0007), Kyiv
  - Odessa Regional Medical Centre of Mental Health (UA0006), Odesa
  - Ukrainian Medical Stomatological Academy, Chair Of Psychiatry, Narcology And Medical Psychology Based On O.F. Maltsev Poltava Regional Clinical Psychiatric Hospital (UA0001), Poltava
  - Vinnitsa National Medical University (UA0002), Vinnitsa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meyer-Lindenberg A, Nielsen J, Such P, Lemming OM, Zambori J, Buller R, der Goltz CV. A double-blind, randomized, placebo-controlled proof of concept study of the efficacy and safety of Lu AF11167 for persistent negative symptoms in people with schizophrenia. Eur Neuropsychopharmacol. 2022 Aug;61:4-14. doi: 10.1016/j.euroneuro.2022.05.009. Epub 2022 Jun 12. PMID 35704951